CLINICAL TRIAL: NCT06377696
Title: Neuro-Oncology Anywhere: Deploying Mayo Clinic's Remote Cognitive Assessment Battery and Wearable Device Monitoring Platform While Assessing the Impact of Metformin on Cognition and Quality of Life in Patients With History of Cranial Radiation
Brief Title: Remote Cognitive Assessment and Wearable Device While Assessing the Impact of Metformin in Patients With History of Cranial Radiation Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MC230713; NCI-2024-02980 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-005512 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-04-16; First posted 2024-04-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Malignant Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Metformin; Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (metformin) (Experimental): Patients receive metformin PO BID for 12 months. Treatment repeats every 28 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients also wear a wearable device to monitor health and undergo neurocognitive test throughout the study.
  Interventions: Other: Medical Device Usage and Evaluation; Drug: Metformin; Other: Neurocognitive Assessment; Other: Questionnaire Administration
- Group B (usual care) (Active Comparator): Patients receive SOC treatment for 12 months. Patients also wear a wearable device to monitor health and undergo neurocognitive test throughout the study.
  Interventions: Other: Best Practice; Other: Medical Device Usage and Evaluation; Other: Neurocognitive Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive SOC
  Other Names: standard of care; standard therapy
  Arms: Group B (usual care)
Other: Medical Device Usage and Evaluation — Wear wearable device
Drug: Metformin — Given PO
  Other Names: N,N-dimethylbiguanide
  Arms: Group A (metformin)
Other: Neurocognitive Assessment — Undergo neurocognitive test
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial evaluates whether patient care can be done remotely for patients having cranial (skull) radiation or who have previously had cranial radiation. In addition, this trial compares study outcomes between patients who get metformin and those who do not. Cranial radiation, an essential component of brain tumor treatment, can result in significant negative effects on cognitive (the ability to clearly think, learn, and remember) function. Wearable devices have been used in the field of neurology for seizure detection and assessment of patients with movement disorders. Wearable device technology has also been implemented for remote monitoring of cancer patients and for cancer clinical trials. Metformin is the active ingredient in a drug used to treat type 2 diabetes mellitus (a condition in which the body cannot control the level of sugar in the blood). It is also being studied in the treatment of cancer. Use of metformin may reduce risk of cognitive decline following radiation therapy within the skull (intracranial). These effects may be further strengthen by addition of device-based physical activity promotion. Mayo Test Drive is a web-based platform for remote self-administered cognitive assessment. Using Mayo Test Drive may help determine whether patient care can be done remotely, while simultaneously evaluating benefits of health promotion through use of a wearable watch device and metformin in preventing radiation-related cognitive decline.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the feasibility of completing serial remote cognitive, activity/sleep, and self-report assessments in clinical trial participants who have previously received cranial radiation.

SECONDARY OBJECTIVES:

I. Assess the acceptance or satisfaction of patients with the remote monitoring in this trial and how these may differ between those who receive metformin versus (vs.) not.

II. Evaluate compliance and feasibility in terms of the adherence to study drug in those randomized to receive metformin.

III. Assess and compare neurocognitive function scores and the impact of receiving metformin + health promotion with wearable device vs. wearable device only.

IV. Assess the safety and tolerability of metformin in patients who have previously received cranial radiation.

EXPLORATORY OBJECTIVES:

I. Investigate the relationship of metformin and other health outcomes such as activity and sleep data and how these compare to the results for patients who are randomized to the control group, who do not receive metformin.

II. Explore potential differences in these compliance and satisfaction measures and how they may correspond to health disparities and social determinants of health.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP A: Patients receive metformin orally (PO) twice day (BID) for 12 months. Treatment repeats every 28 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients also wear a wearable device to monitor health and undergo neurocognitive test throughout the study.

GROUP B: Patients receive standard of care (SOC) treatment for 12 months. Patients also wear a wearable device to monitor health and undergo neurocognitive test throughout the study.

Upon completion of study treatment, patients are followed up at 30 days then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of brain tumor requiring cranial radiation treatment NOTE: Patient may be enrolled during or up to 5 years after completion of cranial radiation administered for treatment of primary or metastatic intracranial tumor
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2, AND Karnofsky performance status (KPS) of ≥ 70
* Expected survival ≥ 6 months in the opinion of treatment team
* Willing and able to adhere with the protocol for the duration of the study including undergoing treatment, and attending scheduled visits, and examinations
* The following laboratory values obtained ≤ 30 days prior to registration:

  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN [≤ 5 x upper limit normal (ULN) for patients with baseline liver disease]
* Negative pregnancy test ≤ 8 days prior to registration for persons of childbearing potential only
* Ability to complete cognitive assessments and questionnaires by themselves or with assistance

Exclusion Criteria:

* Uncontrolled and/or intercurrent illness or other condition which limits safety of or compliance with study proceedings
* Pregnant or nursing, imprisoned, or lacking capacity for understanding
* Unable to swallow tablets or at risk for impaired absorption of oral medication
* Currently taking the study agent (i.e., metformin), and cannot safely discontinue if randomized to the control group (Group B)
* Known hypersensitivity or allergy to metformin
* Current use of resveratrol, CoQ10 (coenzyme Q10), coconut oil/other medium chain triglyceride-containing (e.g., Axona) supplements, or curcumin and unwilling to discontinue prior to registration and remain off these agents for study duration
* Unable to read and speak English. Note: English doses not to need to be primary language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Compliance of patients who complete the testing schedule for the cognitive assessments (Feasibility) | Baseline, 3 months, and 6 months
  Feasibility will be assessed based on compliance of patients to the testing schedule for the cognitive assessments using the Mayo Test Drive tool.

SECONDARY OUTCOMES:
Overall completion rates and compliance (Feasibility) | Up to 12 months
  Will evaluate compliance of completing the patient-reported symptom assessments and the activity and sleep assessments and will assess for any patterns within and between the treatment arms.
Overall satisfaction | Up to 12 months
  Satisfaction/acceptance rates will be evaluated using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C-30, which consists of 30 questions, each answered on a 4-point (e.g., not at all, a little, quite a bit, very much) or a scale of 1-7 where 1=very poor and 7=excellent.
Adherence (Feasibility) | Up to 12 months
  Adherence to study drug will be evaluated in those randomized to the metformin treatment group. Will consider sufficient adherence to be defined as taking at least 80% of the prescribed doses.
Neurocognitive scores | Up to 12 months
  Neurocognitive scores will be assessed using the Mayo Test Drive, a web-based platform for remote self-administered cognitive assessment that uses the Stricker Learning Span (SLS), which is a computer adaptive word-list memory test that matches test difficulty to user performance, and the Symbols test, which is a measure of processing speed and executive functioning that requires timed visual matching. The primary outcome measure will be the Mayo Test Drive raw composite (range 0 - 158). Higher scores indicate better cognitive test performance. Several secondary outcome measures will also be analyzed including but not limited to SLS sum of trials (0-108), an accuracy-weighted Symbols score (0-50), and Symbols average response time for correct items (0+). Participants will have opportunity to provide comments about the testing experience.
Incidence of adverse events (AEs) | Up to 2 years
  Safety and tolerability will be assessed on those randomized to receive metformin, as defined using the Common Terminology Criteria for Adverse Events version 5. Any AEs will be summarized with the maximum grade of each AE reported for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Ugur T. Sener, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials